CLINICAL TRIAL: NCT07049393
Title: Role of Emergency Transport Systems in Improving Cardiac and Respiratory Complications in Road Traffic Accident Cases: A District Level Investigation
Brief Title: Role of ETS in Improving Cardiac and Respiratory Complications in Road Traffic Accident Cases
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/914
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Accident, Traffic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Road traffic accident (RTA) victims(SAQ) — Road traffic accident (RTA) victims present with respiratory and/or cardiac complications. a self-administered questionnaire.
  Patients transported to healthcare facilities in District Karak using emergency transport systems.Road traffic accident (RTA) victims presenting with respiratory and/or cardiac complications.

SUMMARY:
This study will be a Cross-Sectional Study The research will be conducted in the Accident & Emergency (A&E) Department and Trauma Center of District Head Quarter (DHQ), Karak.

Road traffic accident (RTA) victims presenting with respiratory and/or cardiac complications.

Patients transported to healthcare facilities in District Karak using emergency transport systems.

Individuals of all ages and genders involved in RTAs. Cases where detailed medical and transport records are available for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Road traffic accident (RTA) victims presenting with respiratory and/or cardiac complications.
* Patients are transported to healthcare facilities in District Karak using emergency transport systems.
* Individuals of all ages and genders involved in RTAs.
* Cases where detailed medical and transport records are available for analysis.

Exclusion Criteria:

* RTA victims without respiratory or cardiac complications.
* Patients transported by means other than emergency transport systems (e.g., private vehicles).
* Cases with incomplete or missing medical and transport data.
* Victims of RTAs occurring outside the geographic boundaries of District Karak.
* Patients who decline to participate in the study or whose guardians refuse consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Road traffic accident (RTA) victims presenting with respiratory and/or cardiac complications.
  Patients transported to healthcare facilities in District Karak using emergency transport systems.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
structured questionnaire for CR | 12 Months
  structured questionnaire Cardiac and Respiratory Complications in Road Traffic Accident Cases 0-50 soring from lowest to worst

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Centers and Hospitals, Karak, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No